CLINICAL TRIAL: NCT05225883
Title: GEnome-wide Association Study in N-methyl-D-Aspartate Receptor and Other autoiMmune Encephalitis.
Brief Title: GWAS in NMDAR Encephalitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 243
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Autoimmune Encephalitis
Keywords: Autoimmune Encephalitis; paraneoplastic neurological syndromes; NMDAr
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood collected at diagnosis time
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune encephalitis and paraneoplastic neurological syndromes: Patients with well-characterized antibodies against onconeural antigens, synaptic or cell-surface antigens
  Interventions: Genetic: GWAS

INTERVENTIONS:
Genetic: GWAS — This is a non-interventional study involving biological samples (DNA). Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL)/NeuroBioTec (including tissue, cells or biological fluids) and genetic analysis for research purposes (e.g. involving genes related to the disease for which the patient was followed). Additionally, patients will be informed about the present study.

SUMMARY:
Autoimmune encephalitis are characterized by the subacute development of memory deficits, altered mental status, and psychiatric symptoms, generally in association with anti-neuronal antibodies. Two main groups of autoimmune encephalitis may be distinguished based on the location of the targeted antigen: 1) Intracellular antigens, in which the antibodies are thought not to be pathogenic, and the disorders are usually strongly associated with cancer, constituting therefore paraneoplastic neurological syndromes; 2) Synaptic proteins and surface receptors, in which the antibodies are pathogenic and the frequency of cancer is variable depending on the antibody and the demographic characteristics of the patient.

Encephalitis with antibodies against N-methy-D-aspartate receptor is the most common autoimmune encephalitis, being even more frequent than infectious etiologies. It is characterized by subacute onset of memory deficits, psychiatric symptoms, speech dysfunction, seizures, movement disorders, decreased level of consciousness, dysautonomia and central hypoventilation. Nearly 50% of women with anti-NMDAR encephalitis have an ovarian teratoma, while associated tumors in elderly patients are usually carcinomas. In contrast, most cases in children and young men are non-paraneoplastic. Recently, herpes-simplex encephalitis has been described as another trigger of NMDAR encephalitis. Conversely, for the vast majority of the non-paraneoplastic autoimmune encephalitis, no acquired triggers have been described so far.

In addition to acquired susceptibility, genetic predisposition may also be important in the pathogenesis of autoimmune encephalitis. The human leukocyte antigen (HLA) is the genetic factor most frequently associated with autoimmune diseases, and it has been already linked to a few autoimmune encephalitis, such as anti-leucine rich glioma inactivated 1 (LGI1), contactin-associated protein-like 2 (CASPR2), IgLON5, and glutamic acid decarboxylase 65 (GAD65) encephalitis. However, no HLA association has been reported for NMDAR encephalitis, suggesting that in this condition, and likely in others, non-HLA loci might be involved in the pathogenesis as well.

Genome-wide association studies (GWAS) are useful tools to identify variants at genomic loci that are associated with complex diseases, and in particular, to detect associations between single-nucleotide polymorphisms (SNPs) and diseases. The aim of the study is to detect genetic variants in NMDAR encephalitis and other autoimmune encephalitis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of well-characterized antibodies in serum or cerebrospinal fluid;
* Clinical picture compatible with the detected antibody based on the literature

Exclusion Criteria:

* Absence of complete clinicobiological data.
* Alternative diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune encephalitis or paraneoplastic neurological syndromes whose samples were sent for analysis at Centre de Référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, for anti-neural antibody study and then stored at the biobank Neurobiotec.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GWAS in autoimmune encephalitis | 24 month after the beginning of study
  Detection of genetic variants (SNPs) in autoimmune encephalitis

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France